CLINICAL TRIAL: NCT06535841
Title: MTX-474-S101: A Phase 1 Randomized, Double-Blind, Dose-Escalating Study to Assess the Safety, Tolerability, and Pharmacokinetics of MTX-474 in Healthy Adults
Brief Title: A First-in-Human Safety Trial of MTX-474
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mediar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MTX-474-S101
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: MTX-474-S101; MTX-474; Healthy Volunteer; MAD; SAD; Adult; Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MTX-474 (Experimental): Biological: MTX-474
  Interventions: Biological: MTX-474
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MTX-474 — MTX-474 is an immunoglobin G1 (IgG1) monoclonal antibody directed against Ephrin B2 that binds to and has demonstrated ability to block phosphorylation of its preferred receptor EphB4. Increased levels of circulating soluble EphrinB2 have been found in patients with systemic sclerosis.
  Arms: MTX-474
Other: Placebo — Matching Placebo - Normal Saline
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to assess the safety, tolerability, and PK of single and multiple ascending doses of MTX-474 administered in healthy adults.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to assess the safety, tolerability, and PK of single and multiple ascending doses of MTX-474 administered in healthy adults.

SAD Portion

The SAD portion of the study will consist of 6 planned dosing cohorts each comprising 8 healthy participants. The starting dose will be 0.125 mg/kg (Cohort 1) with subsequent planned doses of 0.25 mg/kg (Cohort 2), 0.5 mg/kg (Cohort 3), 1 mg/kg (Cohort 4), 2 mg/kg (Cohort 5), and 4 mg/kg (Cohort 6). Planned doses may be adjusted in response to the data. Additional participants and/or additional dosing cohorts may be added as needed based on the data.

Within each cohort, participants will be randomly assigned to receive MTX-474 or matched placebo. The first 2 participants (sentinel participants) within each cohort will be randomized 1:1 to receive MTX-474 or placebo on Day 1. These participants will be monitored for 24 hours, and after review of the safety data from both participants and approval by the study Investigator, the additional 6 participants will be randomized to study drug (n=5 MTX-474; n=1 placebo).

Each participant will undergo assessments at specified timepoints on Days 1 through 29. End-of-Study (EOS) procedures will be completed on Day 29 or upon early termination (ET). An End-of-Follow-up (EOF) assessment of PK and ADA will be completed on Day 29.

MAD Portion

The MAD portion of the study will consist of 4 planned dosing cohorts. Each cohort will comprise 8 healthy participants (n=6 MTX-474; n=2 placebo). The starting dose will be 0.5 mg/kg (Cohort 1) with subsequent planned doses of 1 mg/kg (Cohort 2), 2 mg/kg (Cohort 3), and 4 mg/kg (Cohort 4). Planned doses may be adjusted in response to the data. Additional participants and/or additional dosing cohorts may be added as needed based on the data.

On Day 1, participants will be randomized to receive either MTX-474 or matched placebo. The randomized participants will receive a dose of study drug on Days 1, 8, 15, and 22. Participants will be housed inpatient from Day -1 through Day 2, Days 7 through 9, 14 through 16, and 21 through 23. All other visits will be conducted in the outpatient setting. Each participant will undergo assessments at specified timepoints on Days 1 through 50. End-of-study procedures will be completed on Day 50, or upon ET. An EOF assessment of PK and ADA will be completed on Day 50.

Safety and tolerability of MTX-474 will be reviewed through Day 29 by the study Investigator and SRMO to inform dose escalation decisions for the next dose cohort.

Additional cohorts for the SAD and MAD portions of the study may be added as needed to potentially explore alternative doses.

ELIGIBILITY:
Inclusion Criteria:

* All genders, ages 18 to 60 years, inclusive
* Willing and able to complete all protocol-required study visits and procedures
* Consumption of not more than 5 cigarettes or other cotinine-containing products (including tobacco, nicotine gum, patches, and e-cigarettes) per week as long as they are willing to abstain nicotine use approximately 5 days prior to admission and during inpatient stays
* Willing to refrain from marijuana- or cannabinol-containing products for 30 days before Screening and until the last study visit
* Agree to a highly effective method of contraception for 28 days prior to the first dose of study drug, and persist through 65 days after the last dose of study drug.

Exclusion Criteria:

* Any concurrent active medical condition determined clinically significant by the Investigator
* Body mass index (BMI) >32 kg/m2 or body weight >100kg
* Use of any systemic immunosuppressant medications, medications to treat diabetes, antipsychotics, anticoagulants, or other medications within 90 days of Screening
* Cancer or a history of cancer or lymphoproliferative disorder within 5 years of Screening other than adequately treated non-melanomatous skin cancers or cervical carcinoma in situ
* Current infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) as evidenced by a positive hepatitis B surface antigen or a positive HIV test at Screening
* Currently pregnant, lactating, or planning to conceive or contribute to pregnancy during the trial and up to 65 days (for women of childbearing potential) or 125 days (for males) after the participant's last dose of study drug, if applicable
* History of severe depression, psychosis, or suicidal ideation within 5 years of Screening
* History of anaphylaxis or other significant allergies in the opinion of the Investigator
* History of substance use disorder as specified in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, within 1 year of Screening
* Positive screen for drugs of abuse or alcohol intake at Screening or admission to the CRU (Day -1)
* Any clinically significant disease or laboratory abnormality detected at Screening that might interfere with a participant's ability to complete the study, on-study evaluations, or participant safety
* Any surgical procedure, including planned procedures within 12 weeks of Screening
* Participation in another research study of an investigational agent within 30 days of Screening or 5 half-lives of the agent, whichever is longer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events in healthy volunteers | Through Day 29 (SAD Cohort) or Day 50 (MAD Cohort)
  Clinical Safety Labs are collected, and Adverse Events are assessed in both inpatient and outpatient clinic visits
MTX-474 PK by dose will be evaluated for Cmax, as feasible | Through Day 29 (SAD Cohort) or Day 50 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study
Serum sample results will be summarized for presence of Anti-Drug Antibodies during the SAD and MAD portions of the study | Through Day 29 (SAD Cohort) or Day 50 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study to assess for the presence and titer (if applicable) of Anti-Drug Antibodies.
MTX-474 PK by dose will be evaluated for AUC0-t, as feasible | Through Day 29 (SAD Cohort) or Day 50 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study
MTX-474 PK by dose will be evaluated for AUC0-tau (MAD only), as feasible | Through Day 29 (SAD Cohort) or Day 50 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study
MTX-474 PK by dose will be evaluated for AUC0-∞, as feasible | Through Day 29 (SAD Cohort) or Day 50 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study

SECONDARY OUTCOMES:
Blood serum samples will be collected to assess the target engagement of MTX-474 in healthy adult participants | Through Day 29 (SAD Cohort) or Day 50 (MAD Cohort)
  These assessments will be summarized as:
  Change from Baseline in bound EphrinB2 levels Change from Baseline in free EphrinB2 levels Change from Baseline in the percent phorphoEphB4 (pEpB4) positive cells and ratio of pEpB4 to total EphB4 positive cells

OTHER OUTCOMES:
To assess the effect of MTX-474 on PD biomarker PRO-C3 for fibrosis in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in fibrosis biomarker PRO-C3 will be evaluated.
To assess the effect of MTX-474 on PD biomarker PRO-C6 for fibrosis in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in fibrosis biomarker PRO-C6 will be evaluated.
To assess the effect of MTX-474 on PD biomarker C7M for fibrosis in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in fibrosis biomarker C7M will be evaluated.
To assess the effect of MTX-474 on PD biomarker PRO-C4 for fibrosis in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in fibrosis biomarker PRO-C4 will be evaluated.
To assess the effect of MTX-474 on PD biomarker IFN-γ for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IFN-γ will be evaluated.
To assess the effect of MTX-474 on PD biomarker IL-1β for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-1β will be evaluated.
To assess the effect of MTX-474 on PD biomarker IL-2 for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-2 will be evaluated.
To assess the effect of MTX-474 on PD biomarker IL-4 for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-4 will be evaluated.
To assess the effect of MTX-474 on PD biomarker IL-6 for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-6 will be evaluated.
To assess the effect of MTX-474 on PD biomarker IL-10 for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-10 will be evaluated.
To assess the effect of MTX-474 on PD biomarker IL-12p70 for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-12p70 will be evaluated.
To assess the effect of MTX-474 on PD biomarker IL-17A for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-17A will be evaluated.
To assess the effect of MTX-474 on PD biomarker TNF-α for inflammation in healthy adult participants | Through Day 50 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker TNF-α will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bornstein, MD, Study Director — Mediar Therapeutics; Gloria Wong, PhD, MBBS, Principal Investigator — Nucleus Network Brisbane
Locations (1):
- Nucleus Network, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No